CLINICAL TRIAL: NCT01644240
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled, Multiple Intravenous Dose Study to Examine the Safety, Tolerability, and Pharmacokinetics of Intravenous TD-8954, a 5-HT4 Receptor Agonist, in Healthy Subjects
Brief Title: A Phase 1, Multiple Intravenous Dose Study to Examine Safety, Tolerability, and PK of Intravenous TD-8954, a 5-HT4 Receptor Agonist, in Healthy Subjects
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: For business reasons
Sponsor: Theravance Biopharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 0095
Record Dates: First submitted 2012-07-13; First posted 2012-07-19 (Estimated); Results first posted 2017-08-02 (Actual); Last update posted 2017-08-02 (Actual); Status verified 2017-04

CONDITIONS: Gastrointestinal Motility Disorder
MeSH Terms: interventions — 4-((4-((2-isopropyl-1H-benzoimidazole-4-carbonyl)amino)methyl)piperidin-1-ylmethyl)piperidine-1-carboxylic acid methyl ester

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- TD-8954 Dose 1 (Experimental)
  Interventions: Drug: TD-8954
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo - saline
- TD-8954 Dose 2 (Experimental)
  Interventions: Drug: TD-8954

INTERVENTIONS:
Drug: TD-8954 — Intravenous infusion
  Arms: TD-8954 Dose 1; TD-8954 Dose 2
Drug: Placebo - saline — Intravenous infusion
  Arms: Placebo

SUMMARY:
This is a single-center, randomized, double-blind, placebo-controlled study to evaluate the safety, tolerability, and pharmacokinetics (PK) of repeated IV doses of TD-8954 in healthy adults 18 to 45 years of age and healthy elderly subjects 65 to 85 years old. A healthy elderly subject population is included to evaluate the safety, tolerability, and PK of TD-8954 IV. Pharmacodynamic effects on bowel movements will also be evaluated. Screening for all cohorts will be conducted within 21 days before the first dose.

ELIGIBILITY:
Inclusion Criteria:

1. For Cohorts 1: adult males and females age 18 to 45 years, inclusive; for Cohorts 2 and 3, adult males and females 65 to 85 years of age, inclusive; for Cohort 4, adult males and females 18 to 45 or 65 to 85 years of age, inclusive.
2. Body mass index (BMI)between 18 to 36 kg/m2, inclusive.
3. Average frequency of ≥ 3 bowel movements per week.

Exclusion Criteria:

1. Persistent symptoms of functional GI disorder (such as irritable bowel syndrome, functional constipation, functional dyspepsia, or other symptom-based GI disorders unexplained by a pathologically based disorder) during the 6 months prior to screening, including a history of major surgery of the GI tract, excluding cholecystectomy and appendectomy.
2. History or presence of clinically significant respiratory, GI, renal, hepatic, endocrine, hematological, neurological (including chronic headache, current or prior psychiatric disease/condition, stroke), cardiovascular, psychiatric, musculoskeletal, genitourinary, immunological, or dermatological disorders. Subjects with mild, chronic, stable disease (e.g., controlled hypertension, controlled hypercholesterolemia, non insulin-dependent diabetes, osteoarthritis) may be enrolled if the condition is well controlled and not anticipated to interfere with the objectives of the study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2012-09 (Actual); Primary Completion 2012-11 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brett Haumann, SVP, Clinical Development, Study Director — Theravance Biopharma, US, Inc.
Locations (1):
- Miami Research Associates, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | TD-8954 Dose 1 | Placebo | TD-8954 Dose 2
Started | 6 | 4 | 6
Completed | 6 | 4 | 6
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | TD-8954 Dose 1 | Placebo | TD-8954 Dose 2 | Total
Number analyzed (Participants) | 6 | 4 | 6 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.2 (4.92) | 37.0 (3.56) | 30.2 (5.98) | 32.6 (5.49)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 3 | 7
  Male | 4 | 2 | 3 | 9
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 6 | 4 | 6 | 16

OUTCOME MEASURES:

1. Primary Outcome: Cmax
Description: Maximum concentration in plasma following dosing on Day 1
Time Frame: Day 1
Population: Sample size was 6 at all time points with the exception of 0.5 hours for dose 2 where value was considered an outlier and one subject was excluded from the PK analysis resulting in sample size of 5.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | TD-8954 Dose 1 | Placebo | TD-8954 Dose 2
Number analyzed (Participants) | 6 | 0 | 5
pg/mL | 6920 (2120) |  | 1200 (275)

2. Primary Outcome: Tmax
Description: Time to maximum plasma concentration
Time Frame: Day 1
Measure: Median (Full Range); unit: hours
Arm/Group | TD-8954 Dose 1 | Placebo | TD-8954 Dose 2
Number analyzed (Participants) | 6 | 0 | 5
hours | 0.983 [0.500 to 0.983] |  | 0.887 [0.500 to 0.983]

3. Primary Outcome: t½
Description: Time to 50% plasma concentration
Time Frame: Day 1
Population: Subjects did not meet extrapolation criteria and were not included in the analysis.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | TD-8954 Dose 1 | Placebo | TD-8954 Dose 2
Number analyzed (Participants) | 3 | 0 | 1
hours | 10.3 (1.22) |  | 8.77

4. Primary Outcome: AUC0-24
Description: Area under the plasma concentration time curve through 24 hours after dosing.
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: pg*hr/mL
Arm/Group | TD-8954 Dose 1 | Placebo | TD-8954 Dose 2
Number analyzed (Participants) | 3 | 0 | 1
pg*hr/mL | 41500 (2740) |  | 12800

5. Primary Outcome: AUC0-∞
Description: Area under the concentration time curve from time 0 to infinity.
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: pg*hr/mL
Arm/Group | TD-8954 Dose 1 | Placebo | TD-8954 Dose 2
Number analyzed (Participants) | 3 | 0 | 1
pg*hr/mL | 50600 (5440) |  | 15300

6. Primary Outcome: AUCtau
Description: Area under the plasma concentration time curve over the dosing interval estimated using the linear trapezoidal rule.
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: pg*hr/mL
Arm/Group | TD-8954 Dose 1 | Placebo | TD-8954 Dose 2
Number analyzed (Participants) | 6 | 0 | 5
pg*hr/mL | 37600 (7070) |  | 8180 (2610)

7. Primary Outcome: Plasma Vz
Description: Volume of distribution
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | TD-8954 Dose 1 | Placebo | TD-8954 Dose 2
Number analyzed (Participants) | 3 | 0 | 1
Liters | 147 (9.37) |  | 82.8

8. Primary Outcome: Plasma CL
Description: Plasma clearance
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: L/hr
Arm/Group | TD-8954 Dose 1 | Placebo | TD-8954 Dose 2
Number analyzed (Participants) | 3 | 0 | 1
L/hr | 9.95 (1.03) |  | 6.55

9. Primary Outcome: Cmax
Description: Maximum plasma concentration
Time Frame: Day 5
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | TD-8954 Dose 1 | Placebo | TD-8954 Dose 2
Number analyzed (Participants) | 6 | 0 | 6
pg/mL | 7070 (1550) |  | 7600 (1650)

10. Secondary Outcome: Number of Subjects With Adverse Events
Time Frame: 1 week
Measure: Number; unit: participants
Arm/Group | TD-8954 Dose 1 | Placebo | TD-8954 Dose 2
Number analyzed (Participants) | 6 | 4 | 6
participants | 5 | 1 | 2

11. Primary Outcome: Tmax
Description: Time to reach maximum plasma concentration.
Time Frame: Day 5
Measure: Median (Full Range); unit: hours
Arm/Group | TD-8954 Dose 1 | Placebo | TD-8954 Dose 2
Number analyzed (Participants) | 6 | 0 | 6
hours | 0.983 [0.500 to 1.02] |  | 0.983 [0.500 to 0.983]

12. Primary Outcome: t½
Description: Time to 50% plasma concentration
Time Frame: Day 5
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | TD-8954 Dose 1 | Placebo | TD-8954 Dose 2
Number analyzed (Participants) | 6 | 0 | 6
hours | 18.0 (3.18) |  | 18.9 (3.47)

13. Primary Outcome: AUC0-24
Description: Area under the plasma concentration time curve 24 hours following the last dose.
Time Frame: Day 5
Measure: Mean (Standard Deviation); unit: pg*hr/mL
Arm/Group | TD-8954 Dose 1 | Placebo | TD-8954 Dose 2
Number analyzed (Participants) | 6 | 0 | 6
pg*hr/mL | 51000 (9310) |  | 63300 (11800)

14. Primary Outcome: AUC0-∞
Description: Area under the plasma concentration time curve from 0 to infinity.
Time Frame: Day 5
Measure: Mean (Standard Deviation); unit: pg*hr/mL
Arm/Group | TD-8954 Dose 1 | Placebo | TD-8954 Dose 2
Number analyzed (Participants) | 6 | 0 | 6
pg*hr/mL | 80400 (15700) |  | 102000 (12300)

15. Primary Outcome: AUCtau
Description: Area under the plasma concentration time curve over the dosing interval estimated using the linear trapezoidal rule.
Time Frame: Day 5
Measure: Mean (Standard Deviation); unit: pg*hr/mL
Arm/Group | TD-8954 Dose 1 | Placebo | TD-8954 Dose 2
Number analyzed (Participants) | 6 | 0 | 6
pg*hr/mL | 68700 (12700) |  | 86300 (12800)

16. Primary Outcome: Vss
Description: Apparent volume of distribution at steady state
Time Frame: Day 5
Measure: Mean (Standard Deviation); unit: L
Arm/Group | TD-8954 Dose 1 | Placebo | TD-8954 Dose 2
Number analyzed (Participants) | 6 | 0 | 6
L | 225 (68.1) |  | 194 (60.4)

17. Primary Outcome: CLss
Description: Apparent clearance
Time Frame: Day 5
Measure: Mean (Standard Deviation); unit: L/hr
Arm/Group | TD-8954 Dose 1 | Placebo | TD-8954 Dose 2
Number analyzed (Participants) | 6 | 0 | 6
L/hr | 10.1 (2.00) |  | 8.11 (1.34)

ADVERSE EVENTS:
Arm/Group | TD-8954 Dose 1 | Placebo | TD-8954 Dose 2
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/4 | 0/6
Other Adverse Events (participants affected / at risk) | 5/6 | 1/4 | 2/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TD-8954 Dose 1 (N=6) | Placebo (N=4) | TD-8954 Dose 2 (N=6)
Headache (Nervous system disorders) | 4 (4) | 0 (0) | 1 (1)
Dizziness Postural (Nervous system disorders) | 2 (2) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Infusion Site Extravasation (General disorders) | 1 (1) | 0 (0) | 0 (0)
Transaminases Increased (Investigations) | 1 (1) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI may communicate the trial results generated by the PI, but only after the first publication or presentation of the combined study results generated by all participating sites. The Sponsor can then review trial results communications prior to public release and can embargo communications regarding trial results for a period that is more than 60 days but less than or equal to 180 days. The Sponsor cannot require changes to the communication and cannot extend the embargo.